CLINICAL TRIAL: NCT07104565
Title: A Phase 2a, Open-Label, Multicenter Study of Tafasitamab in Adult Participants With Primary Autoimmune Blood Cell Disorders
Brief Title: Study to Assess the Safety and Tolerability of Tafasitamab in Adult Participants With Primary Autoimmune Blood Cell Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA000585-201
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenia
Keywords: primary warm autoimmune hemolytic anemia; primary immune thrombocytopenia; anti-CD19 monoclonal antibody
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - primary immune thrombocytopenia (ITP) (Experimental): INCA000585 will be administered intravenously.
  Interventions: Drug: INCA000585
- Cohort 2 - primary warm autoimmune hemolytic anemia (wAIHA) (Experimental): INCA000585 will be administered intravenously.
  Interventions: Drug: INCA000585

INTERVENTIONS:
Drug: INCA000585 — Tafasitamab will be administered intravenously at protocol defined timepoints.

SUMMARY:
This study will evaluate the safety and efficacy of tafasitamab in adult participants with primary autoimmune blood cell disorders.

ELIGIBILITY:
Inclusion Criteria:

- Ability to comprehend and willingness to sign a written ICF for the study.

* Aged ≥ 18 years.
* Confirmed historical diagnosis of one of the following autoimmune blood disorders:

  * Primary ITP.
  * Primary wAIHA.
* No history of splenectomy.
* Confirmed transient response to at least 1 prior early-line treatment (eg, corticosteroids, IVIG, rituximab):

  * Primary ITP: Increase in platelet count to ≥ 30 × 109/L with at least a 2-fold increase of baseline platelet count.
  * Primary wAIHA: Increase in hemoglobin to ≥ 10 g/dL with an increase of at least 2 g/dL from baseline.
* Received ≥ 1 standard course of rituximab (375 mg/kg × 4 weekly doses or 2 doses of 1000 mg flat dose every 2 weeks) with last dose given at least 6 months prior to initiation of study treatment. Note: If rituximab was the only prior therapy, individuals with NR to rituximab will not be eligible.

  * Primary ITP: a PR (platelet count ≥ 30 × 109/L with at least a 2-fold increase of baseline platelet count) within 6 months of the last administered dose followed by relapse OR a CR (platelet count > 100 × 109/L) lasting < 48 weeks OR NR (platelet count < 30 × 109/L or less than 2-fold increase of baseline platelet count or bleeding) within 6 months of the last administered dose.
  * Primary wAIHA: a PR with hemoglobin ≥ 10 g/dL and with an increase of at least 2 g/dL from baseline OR a CR (hemoglobin ≥ 12 g/dL and normalization of hemolytic markers) OR NR (hemoglobin < 10 g/dL or < 2 g/dL increase of baseline hemoglobin).
* Persistent or chronic active primary ITP or active primary wAIHA with indication for treatment at the time of inclusion.

  * Primary ITP: platelet count < 30 × 109/L within the 15 days before treatment is scheduled to begin (Day 1).

Note: Participants treated with a rescue therapy during screening in response to a documented platelet count < 30 × 109/L are eligible, irrespective of platelet count within 15 days of Day 1.

• Primary wAIHA: hemoglobin < 10 g/dL documented with DAT result positive for IgG, with or without C3d, and evidence of hemolysis based on low haptoglobin, elevated LDH, and/or indirect bilirubin.

* ECOG performance status of 0 to 2.
* Willingness to avoid pregnancy or fathering children.
* Further inclusion criteria apply.

Exclusion Criteria:

* Clinical manifestations typical for cold agglutinin disease.
* Life-threatening bleeding or urgent need to elevate the platelet count for primary ITP or hemodynamic instability or hemoglobin < 6 g/dL with urgent need to elevate hemoglobin for primary wAIHA within 2 weeks prior to Day 1.
* Prior treatment with anti-CD19 therapy (eg, mAb, bispecific T-cell engager, or CAR T cell) for any indication.
* Previous severe allergic reaction to a mAb or known allergy to any component/excipient of tafasitamab.
* Changes in doses (> 10%) of permitted disease-related therapies, including oral corticosteroids and TPO-RA (primary ITP participants) within 2 weeks prior to Day 1, or change in ESA (primary wAIHA participants) dose within 2 weeks prior to Day 1.
* Evidence of hypogammaglobulinemia during screening (IgA < 70 mg/dL, IgG < 700 mg/dL, and/or IgM < 40 mg/dL) and frequent and/or severe infections.
* Women who are pregnant or breastfeeding.
* History of malignancy except for the following:

  * Malignancy treated with curative intent with no evidence of active disease for more than 2 years before screening.
  * Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanoma skin cancer.
  * Adequately treated carcinoma in situ without current evidence of disease.
* Congestive heart failure (left ventricular ejection fraction of < 50%, assessed by 2 dimensional echocardiography or a multigated acquisition scan).
* Participants with:

  * Known positive test result for HCV (with HCV antibody serology testing) and a positive test for HCV RNA.

Note: Participants with positive serology must have been tested for HCV RNA and are eligible only in the case of negative HCV RNA test result.

• Known positive test result for chronic HBV infection (defined by HBsAg positivity or positive HBV DNA test result).

Note: Participants with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA was undetectable, provided that they are willing to undergo monthly ongoing DNA testing. Antiviral prophylaxis may be administered as per institutional guidelines.

Note: Participants who have protective titers of HBsAb (HBsAb positive, HBcAb negative, and HBsAg negative) after vaccination or prior HBV infection are eligible.

• Seropositivity for or history of active viral infection with HIV.

* Active systemic infection (including infection with SARS-CoV-2).
* Participants in a severely immunocompromised state, per investigator's clinical assessment.
* Receipt of a live-attenuated vaccine within 4 weeks prior to the first infusion of tafasitamab (inactivated and killed vaccines are acceptable).
* Coagulation or platelet function abnormality.
* An active medical condition with a strong indication for treatment with anticoagulation agents (eg, intracoronary stent within 12 months).
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Toxicities related to prior therapies must be CTCAE (v5.0) ≤ Grade 1 at the time of study treatment/enrollment (except for chronic toxicities [≤ Grade 2] not expected to resolve).
* Chronic infectious disease requiring systemic antibiotics or antifungal or antiviral medications.
* Unwillingness to undergo transfusion with blood components.
* Current use of prohibited medication as described in the protocol.
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 52 weeks
  Defined as any adverse event, either reported for the first time or worsening of a pre-existing event after the first dose of study drug up to 90 days after the last dose of study drug.
Stable platelet response | After Day 56 up to Week 48
  Defined as platelet count ≥ 50 × 109/L in the absence of clinically significant bleeding or rescue therapy at ≥ 2 consecutive assessments any time after Day 56 until Week 48 in participants with primary ITP.
Stable hemoglobin response | After Day 56 up to Week 48
  Defined as hemoglobin ≥ 10 g/dL and a ≥ 2 g/dL increase from baseline in the absence of rescue therapy at ≥ 2 consecutive assessments any time after Day 56 until Week 48 in participants with primary wAIHA.

SECONDARY OUTCOMES:
Complete Response (CR) | Week 24
  Defined as platelet count ≥ 100 × 109/L at Week 24 in the absence of clinically significant bleeding or rescue therapy in participants with primary ITP.
CR (complete remission) | Week 48
  Defined as platelet count ≥ 100 × 109/L at Week 48 in the absence of clinically significant bleeding or rescue therapy in participants with primary ITP.
Partial Response (PR) | Week 24
  Defined as platelet count ≥ 30 × 109/L and at least a 2-fold increase of baseline platelet count at Week 24 in the absence of clinically significant bleeding or rescue therapy in participants with primary ITP.
Duration of stable platelet response | Up to Week 48
  Defined as time from start of stable platelet response to loss of platelet response (< 50 × 109/L), clinically significant bleeding, need for rescue therapy, or death, whichever occurs first in participants with primary ITP.
Duration of CR | Up to Week 48
  Defined as time from the start of CR to loss of CR (platelet count < 100 × 109/L), clinically significant bleeding, need for rescue therapy, or death, whichever occurs first in participants with primary ITP.
Duration of response | Up to Week 48
  Defined as time from the date of the first response (PR or CR) to the loss of response (platelet count < 30 × 109/L or a less than a 2-fold increase of baseline platelet count), clinically significant bleeding, need for rescue therapy, or death, whichever occurs first in participants with primary ITP.
CR | Week 24
  Defined as hemoglobin ≥ 12 g/dL and normalization of hemolytic markers (unconjugated bilirubin, LDH, haptoglobin, and reticulocytes) at Week 24 in the absence of rescue therapy in participants with primary wAIHA.
CR (Complete remission) | Week 48
  Defined as hemoglobin ≥ 12 g/dL and normalization of hemolytic markers (unconjugated bilirubin, LDH, haptoglobin, and reticulocytes) at Week 48 in the absence of rescue therapy in participants with primary wAIHA.
PR | Week 24
  Defined as hemoglobin ≥ 10 g/dL and a ≥ 2 g/dL increase from baseline at Week 24 in the absence of rescue therapy in participants with primary wAIHA.
Duration of stable hemoglobin response | Up to Week 48
  Defined as time from start of stable hemoglobin response to loss of stable hemoglobin response (< 10 g/dL or a < 2 g/dL increase from baseline), need for rescue therapy, or death, whichever occurs first in participants with primary wAIHA.
Duration of CR | Up to Week 48
  Defined as time from start of CR to loss of CR (hemoglobin < 12 g/dL or abnormal hemolytic markers [unconjugated bilirubin, LDH, haptoglobin, and reticulocytes]), need for rescue therapy, or death, whichever occurs first in participants with primary wAIHA.
Duration of response | Up to Week 48
  Defined as time from the date of the first response (PR or CR) to the loss of response (hemoglobin < 10 g/dL), need for rescue therapy, or death, whichever occurs first in participants with primary wAIHA.
Serum concentrations of tafasitamab | Up to Week 48
  Serum concentrations of tafasitamab at each assessed timepoint.
Change from baseline in serum antidrug antibody levels | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (39):
- United States (9):
  - Palo Verde Cancer Specialists Palo Verde Hematology Oncology, Ltd Glendale, Glendale, Arizona
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Gnp Research, Cooper City, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Versiti Bloodcenter of Wisconsin Bcw Milwaukee, Milwaukee, Wisconsin
- Australia (6):
  - St Vincent'S Hospital Sydney, Darlinghurst, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre Clayton, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- France (7):
  - Chu Angers - Hôpital Hôtel Dieu, Angers
  - Chu Caen - Hôpital de La Côte de Nacre, Caen
  - Hôpital Henri Mondor, Créteil
  - Chu Dijon - Hopital Du Bocage, Dijon
  - Chu Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Hopital Purpan, Toulouse
  - Chru de Nancy- Hopital de Brabois, Vandœuvre-lès-Nancy
- Italy (8):
  - Azienda Ospedaliero-Universitaria Orsola-Malpighi - Universita Degli Studi Di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia (Presidio Montichiari), Brescia
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Fondazione Irccs Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico Ii, Napoli
  - Azienda Ospedale Universita Di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
- Netherlands (4):
  - Amsterdam Umc, Locatie Vumc, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Spain (2):
  - Ico Badalona - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario La Paz, Madrid
- United Kingdom (3):
  - Castle Hill Hospital, Cottingham
  - Barts Hospital, London
  - Plymouth Hospitals Nhs Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Study to Assess the Safety and Tolerability of Tafasitamab in Adult Participants With Primary Autoimmune Blood Cell Disorders — https://incyteclinicaltrials.com/studies/inca000585-201